CLINICAL TRIAL: NCT00220103
Title: Pre-operative Epirubicin, Capecitabine (Xeloda) and Cisplatin in Patients With Newly Diagnosed Localised Oesophageal Adenocarcinoma
Brief Title: Pre-operative Epirubicin, Cisplatin, and Capecitabine in Patients With Newly Diagnosed Localised Oesophageal Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Jane Lawrence, Royal Marsden NHS Foundation Trust
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2185
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2009-12-16 (Estimated); Status verified 2009-12

CONDITIONS: Adenocarcinoma of Oesophagus
MeSH Terms: conditions — Adenocarcinoma Of Esophagus | interventions — Epirubicin; Capecitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: epirubicin, capecitabine, cisplatin
Procedure: Surgical resection

SUMMARY:
To investigate the efficacy and safety of epirubicin, cisplatin and capecitabine as neoadjuvant therapy prior to radical resection in patients with newly diagnosed operable oesophageal adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Histologically verified adenocarcinoma of the thoracic oesophagus or type 1, 2 and 3 tumours of the oesophagogastric junction (type 1 refers to lower oesophageal, type 2 refers to cardial and type 3 refers to subcardinal cancers).
* AJCC Stage II-III (T2-3 N0-1 M0) (28), as assessed by spiral or multi-slice CT and endoscopic ultrasound, where primary surgery would be considered with curative intent.
* No previous chemotherapy, radiotherapy or other investigational drug treatment for this indication.
* WHO performance status 0,1 or 2.
* Adequate bone marrow function with platelets > 100 x 109/l; WBC > 3 x 109/l; neutrophils > 1.5 x 109/l at the time of study entry.
* Serum bilirubin < 35 mol/l.
* Serum creatinine < 180 mol/l and measured creatinine clearance over 60ml/min.
* No concurrent uncontrolled medical condition.
* No previous malignant disease other than non-melanotic skin cancer or carcinoma in situ of the uterine cervix in the last 10 years.
* Life expectancy > 3 months.
* Adequate contraceptive precautions if relevant.
* Informed written consent.

Exclusion Criteria:

* The presence of locally advanced or metastatic disease precluding curative surgical resection (T4 or Stage IV or M1a-b)
* Total dysphagia (O'Rourke's swallowing function scoring system 5) precluding swallowing of capecitabine even when crushed
* Medical or psychiatric conditions that compromise the patient's ability to give informed consent.
* Patients with disease in any of the following areas on the basis of CT scan and/or endoscopic ultrasound:

  * Evidence of liver, lung or other distant metastases
  * Para-aortic/coeliac lymphadenopathy > 1cm diameter on CT, > 6mm diameter on EUS
  * Invasion of airways, aorta, pericardium, or lung
* New York Heart Association classification Grade III or IV.
* Uncontrolled angina pectoris.
* Pregnancy or breast feeding.
* Impaired renal function with measured creatinine clearance less than 60 ml/min.
* Known malabsorption syndromes.
* Patients with a known hypersensitivity to 5-FU or with a dihydropyrimidine dehydrogenase (DPD) deficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2002-11

PRIMARY OUTCOMES:
Pathological complete response rate

SECONDARY OUTCOMES:
Progression free survival
Overall survival
Objective response rate assessed by CT and EUS
Treatment related toxicity including peri-operative complications
Time to improvement of dysphagia
Pattern of treatment failure
To assess the value of high resolution MRI to depict response to treatment and compare it with EUS and histopathology

CONTACTS AND LOCATIONS:
Overall Officials: David Cunningham, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom